CLINICAL TRIAL: NCT02050971
Title: Safety and Effectiveness Phase 1 Study of Autologous Umbilical Cord Blood Transfusion for the Prevention and Treatment of Prematurity Complications In Preterm Neonates
Brief Title: Autologous Cord Blood Infusion for the Prevention and Treatment of Prematurity Complications In Preterm Neonates
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Milosz Kawa, Boguslaw Machalinski, Professor and Chief, Department of General Pathology, Pomeranian Medical University, Pomeranian Medical University Szczecin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZPO 01; CB-P#1 (Other: Department of General Pathology of PMU)
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Anemia, Neonatal; Intracranial Hemorrhages; Necrotizing Enterocolitis; Respiratory Distress Syndrome, Newborn; Retinopathy of Prematurity; Bronchopulmonary Dysplasia
Keywords: Umbilical Cord Blood; Autologous Umbilical Cord Blood Transfusion; Prematurity Complications; Infant, Premature, Diseases; Infant, Newborn, Diseases; Hematologic Diseases; Lung Diseases; Central Nervous System Diseases; Gastrointestinal Tract Diseases; Vascular Diseases; Retinopathies, Neonates; Prevention,Treatment
MeSH Terms: conditions — Anemia, Neonatal; Intracranial Hemorrhages; Enterocolitis, Necrotizing; Respiratory Distress Syndrome, Newborn; Retinopathy of Prematurity; Bronchopulmonary Dysplasia; Infant, Premature, Diseases; Infant, Newborn, Diseases; Hematologic Diseases; Lung Diseases; Central Nervous System Diseases; Vascular Diseases; Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous cord blood transfusion (Active Comparator): Treatment Group 1 Interventions: collected autologous whole cord blood at birth will be transfused for the preterm neonate
  Interventions: Biological: Umbilical Cord Blood Infusion
- Standard treatment for neonatal anemia (Sham Comparator): Treatment Group 2 Interventions: transfusion of allogeneic whole peripheral blood or any of its components at a time of anemia of prematurity development
  Interventions: Biological: Intravenous Infusion of Peripheral Blood or its Components

INTERVENTIONS:
Biological: Umbilical Cord Blood Infusion — Cord blood collection after delivery of the baby. Preservation of blood in blood bank. Transfusion of autologous cord blood within the first 5 postnatal days.
  Other Names: Whole Autologous Umbilical Cord Blood Infusion
  Arms: Autologous cord blood transfusion
Biological: Intravenous Infusion of Peripheral Blood or its Components — Regular treatment of neonatal anemia with peripheral blood or its components transfusion.
  Other Names: Allogeneic peripheral blood or its components transfusion
  Arms: Standard treatment for neonatal anemia

SUMMARY:
The purpose of this study is to test the safety and effectiveness of a whole own (autologous) umbilical cord blood transfusion in the first 5 days after birth if the baby is born premature <34 weeks and developed anemia of prematurity.

DETAILED DESCRIPTION:
The purpose of this pilot study is to conduct the investigation of the safety and efficacy of autologous cord blood infusion in premature neonates who demonstrate anemia due to prematurity (most common prematurity complication). However, premature infants reveal a high risk of other acute complications, including brain injury (e.g., intraventricular hemorrhage; IVH), necrotizing enterocolitis (NEC), and neonatal respiratory distress syndrome (RDS), as well as retinopathy of prematurity (ROP) and bronchopulmonary dysplasia (BPD). Therefore, prematurity is considered one of the main causes of neonatal deaths. The preterm neonates need transfusion of allogenic whole peripheral blood or any of its components at a time of anemia of prematurity development. In contrast, other prematurity complications do not have effective treatment nor preventive strategies. We will enroll premature neonates born premature (<34 weeks of gestation) who developed anemia of prematurity and had their own autologous cord blood collected for subsequent transfusion. Next, we will test tolerability, safety and efficacy of autogenic whole cord blood infusion and evaluate the frequency of premature complications in neonates after transfusion. Besides, this pilot study will test feasibility of technical collection, preparation and infusion of a neonate's own umbilical cord blood within the first 5 days after birth.

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates less than 34 weeks of gestation, who developed anemia of prematurity,
* available unit of autologous umbilical cord blood

Exclusion Criteria:

* major congenital or chromosomal abnormalities,
* intrauterine infection,
* cyanotic heart defect,
* chronic intrauterine hypoxia (defined as growth retardation or pathologies of placental perfusion),
* incompatibilities in main blood groups and Rh antygen,
* lack of parental consent for enrollment to the study,
* contraindications for cord blood collection (lack of consent, amniotic fluid leakage for longer than 6 hours or physical complications in the cord blood harvesting).

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Safety of autologous cord blood infusion in enrolled preterm neonates. | 1 year
  Confirm the safety of autologous cord blood infusion in preterm neonates by repeated follow-up over one year with clinical and laboratory evaluations.

SECONDARY OUTCOMES:
Efficacy of autologous cord blood infusion in enrolled preterm neonates. | 1 year
  Confirm the efficacy of autologous cord blood infusion in preterm neonates by repeated follow-up over one year with clinical and laboratory evaluations for neurodevelopmental and general health outcomes at 3, 6 and 12 months of age. Particularly, analysis of prematurity complications will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Boguslaw Machalinski, MD, PhD, BSc, Study Chair — Department of General Pathology, Pomeranian Medical University in Szczecin, Poland; Jacek Rudnicki, MD, PhD, BSc, Study Director — Department of Neonatology, Pomeranian Medical University in Szczecin, Poland; Milosz Piotr Kawa, MD, PhD, Principal Investigator — Department of General Pathology, Pomeranian Medical University in Szczecin, Poland
Locations (1):
- Department of Neonatology of Pomeranian Medical University in Szczecin, Poland, Szczecin, Poland

REFERENCES:
- [Derived] Rudnicki J, Kawa MP, Kotowski M, Michalczyk B, Ustianowski P, Czajka R, Machalinski B. Clinical Evaluation of the Safety and Feasibility of Whole Autologous Cord Blood Transplant as a Source of Stem and Progenitor Cells for Extremely Premature Neonates: Preliminary Report. Exp Clin Transplant. 2015 Dec;13(6):563-72. PMID 26643677
- See also: Website of the Pomeranian Medical University in Szczecin, Poland — http://www.pum.edu.pl